CLINICAL TRIAL: NCT04538755
Title: Effect of DAW2020 on Endotypic Traits in OSA
Brief Title: DAW2020 on OSA Endotypic Traits
Acronym: SedOSA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020p002760-1
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule 4 hours before sleep
  Interventions: Drug: Placebo oral capsule
- DAW2020 (Active Comparator): DAW2020 capsule 4 hours before sleep
  Interventions: Drug: DAW2020 oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo before sleep
  Arms: Placebo
Drug: DAW2020 oral capsule — DAW2020 34 mg 4 h before sleep, single night administration
  Arms: DAW2020

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. Some OSA patients with low arousal threshold wake up prematurely during an obstructive event and do not have time for spontaneous upper airway (UA) dilator muscle recruitment. As a consequence they are exposed to apnea and hypopnea cycling. In this protocol the investigators will test the effect of DAW2020 administered before sleep on OSA phenotype traits and OSA severity during sleep.

DETAILED DESCRIPTION:
Two overnight sleep studies will be performed: a drug night and a placebo night. The patient will breath spontaneously (without CPAP) for both nights. On the study nights, subjects will present to the laboratory in the evening and be instrumented with a full polysomnigraphy for monitoring sleep, physiological variables (endotypes), and respiratory events. A history and physical examination will be performed on each night prior to beginning the study, as will a urine pregnancy test in premenopausal women. DAW2020 34 mg will be given 4 hours before lights out. Subjects will sleep at least 50% of the night in the supine position. At least four hours of sleep with high quality signal acquisition will be required for a study to be judged adequate. After the first overnight study is completed, there will be a one-week washout period prior to crossing over to the other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe OSA (AHI ≥ 15 events/hr)

Exclusion Criteria:

* All participants will be healthy and without major organ system disease that would preclude undergoing the physiological measurements.
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, acetazolamide, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Use of SNRIs/SSRIs.
* Conditions likely to affect OSA physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Sleep disordered breathing or respiratory disorders other than obstructive sleep apnea:
* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Hypersensitivity to the study drug (angioedema or urticaria)
* Contraindications to DAW2020
* Use of medications that lengthen QTc interval
* Hypokaliemia, hypomagnesemia, uncontrolled thyroid disease
* Severe claustrophobia.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Effects of DAW2020 on arousal threshold (%eupnea) | 1 night
  Arousal threshold will be calculated using diaphragm EMG

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messineo L, Gell L, Calianese N, Sofer T, Vena D, Azarbarzin A, Labarca G, Taranto-Montemurro L, Yang HC, Wang TY, Kim M, Smith H, White D, Sands S, Wellman A. Effect of Pimavanserin on the Respiratory Arousal Threshold from Sleep: A Randomized Trial. Ann Am Thorac Soc. 2022 Dec;19(12):2062-2069. doi: 10.1513/AnnalsATS.202205-419OC. PMID 35947827